CLINICAL TRIAL: NCT03304743
Title: Dental Panoramic Radiographs to Screen for Post-menopausal Osteoporosis
Acronym: OsteoPano
Status: Completed | Type: Observational
Sponsor: University of Parma (Other)
Collaborators: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Dr Elena Calciolari, Dr, MS, Phd, Clinical Research Fellow, University of Parma
Other Study IDs: P-001
Record Dates: First submitted 2017-09-21; First posted 2017-10-09 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: dental panoramic radiographs; osteoporosis; feasibility study
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-menopausal women: A cohort of 124 consecutive post-menopausal women that performed a DXA scan within the previous 12 months
  Interventions: Diagnostic Test: Dental panoramic radiograph

INTERVENTIONS:
Diagnostic Test: Dental panoramic radiograph — If not performed within the previous 12 months at the Centre of Dentistry, an OPG will be performed during enrolment visit.
  OPGs are routine low-dose x-rays that are often performed during dental check-ups, follow-ups or before dental treatments (e.g. extractions, implant placement, etc.), as they allow the evaluation of both bone and dental structures of both jaws, the sinus and temporo-mandibular joints.

SUMMARY:
Osteoporosis is a common disease that makes the bones fragile and easy to break. Osteoporotic fractures are a serious health problem resulting in pain, reduced mobility, increasing degree of dependence and sometimes death.

Osteoporosis is currently diagnosed by measuring bone density at the hip/spine through an exam called DXA. Although all post-menopausal women are at higher risk, currently Italian national guidelines do not recommend population-screening programs. This leads to several cases not being identified before a fracture occurs.

Since dental panoramic radiographs (OPGs) are common procedures during dental check-ups or before dental treatments, it would be of great value if dentists could use them to identify people with unknown osteoporosis and early refer them to a specialist before they fracture.

While several studies support the use of panoramic indices, they have never been tested in an Italian University Hospital setting and in a study adequately powered and controlled for confounding variables.

The aim of this study is to assess the feasibility of using dental panoramic indices to screen for post-menopausal osteoporosis.

DETAILED DESCRIPTION:
Background:

The World Health Organization (WHO) has defined osteoporosis as a level of bone mineral density (BMD), calculated with DXA (Dual-energy X-ray absorptiometry) technique, 2.5 standard deviations (SD) or more below the average mean value of young healthy women (T-score ≤ -2.5) (Kanis et al., 2013).

Although the WHO reports that there is indirect evidence supporting screening programs in women aged 65 or older, current Italian national guidelines do not recommend population-screening programs for osteoporosis (SIOMMMS 2015). As a consequence, a significant part of Italian osteoporotic patients that may develop a fracture is left undetected and untreated. Although it is recommended to assess risk of osteoporotic fractures with the WHO FRAX tool in all women ≥65 years and men ≥75 years and refer for DXA accordingly, it is not clear how well this tool has been adopted by general practitioners (GPs) in Italy.

Considering the high percentage of people attending regular dental visits (> 22 million according to ISTAT 2013) and the fact that panoramic radiographs of the jawbones are a common procedure that is performed during routine dental check-ups or before several dental treatments, it could be of great clinical value if dentists could opportunistically use panoramic X-rays to identify patients at a high risk of osteoporosis.

In the past years, specific quantitative and qualitative indices/parameters, which can be calculated on dental panoramic radiographs, have been proposed as tools to detect osteoporosis, with different levels of accuracy.

Amongst the quantitative indices, the most adopted ones are the mandibular cortical width (MCW) and the panoramic mandibular index (PMI). The MCW represents the width of the mandibular cortex and it is measured in the mental foramen region, along a line passing through the middle of the mental foramen and perpendicular to the tangent to the lower border of the mandible. The PMI represents the ratio between the mandibular cortical width at mental foramen region and the distance from the lower border to the inferior edge of the mental foramen.

Amongst the qualitative indices, the Klemetti index (KI) is by far the most applied one. KI qualitatively classifies the mandibular cortex distally to the mental foramen in the following categories: C1, when the endosteal margin is even and sharp; C2, when the endosteal margin presents lacunar resorption or cortical residues on one or both sides; and C3, when the cortical layer is clearly porous, with heavy endosteal cortical residues. A recent systematic review and meta-analysis from our group showed that the presence of any kind of cortical porosity (C2+C3) is associated to a sensitivity and specificity in detecting osteoporosis of 80.6% and 64.3%, respectively. The advantage of using this index, compared to other available indices, is that it is straightforward and relatively easy to measure and it does not require specific softwares.

It is clear that the panoramic indices cannot replace the diagnosis of osteoporosis by BMD measurement with DXA scan. However, whenever a panoramic radiograph is available, they might be opportunistically used to detect previously undiagnosed osteoporotic patients and refer them to a specialist before they develop a fracture.

While several studies support the use of panoramic indices, they have never been tested in an Italian University Hospital setting and in a study adequately powered and controlled for confounding variables.

Study description:

This is cross-sectional observational study aiming to recruit a cohort of 124 consecutive post-menopausal women. The only study visit will take place at the "Centro Universitario di Odontoiatria, Dipartimento di Medicina e Chirurgia, Università di Parma".

All post-menopausal women ≥ 65 years old attending the Centro Universitario di Odontoiatria in the new patients' or follow-ups' clinics will be approached to check for the inclusion/exclusion criteria and their willingness to take part in the study. Furthermore, doctors (general practitioners or osteoporosis specialists) will be contacted and will be kindly asked to inform their patient that had done a DXA scan within the past 12 months about the study. Potentially eligible patients will be booked an appointment at the "Centro Universitario di Odontoiatria, Dipartimento di Medicina e Chirurgia, Università di Parma" to check for inclusion/exclusion criteria and for the recruitment. As part of the study, they will receive a full-mouth examination of the hard and soft tissues and an OPG at no cost.

Only 1 study visit will be performed.

Visit 1 (Data collection)

* Signing of informed consent;
* Recording of any concomitant medication;
* Confirmation of participant eligibility in relation to the inclusion/exclusion criteria;
* Examination of hard and soft tissues;
* Full-mouth six-points periodontal chart, with recording of probing pocket depth (PPD), recession (REC), furcation involvement and mobility.
* Dental panoramic radiograph (OPG) if not performed at the Centro Universitario di Odontoiatria within the previous 12 months

Photos of the teeth may be taken to facilitate case documentation. Subjects will not be identifiable.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 years old
* In self-reported menopause, defined as the permanent cessation of ovulation, for at least one year (Soules et al., 2001).
* With a DXA examination at the hip and lumbar spine performed within the previous 12 months

Exclusion Criteria:

* Affected by systemic diseases (with the exception of osteoporosis) recognized to severely affect bone metabolism (e.g. Cushing's syndrome, Addison's disease, diabetes mellitus type 1, leukaemia, pernicious anaemia, malabsorption syndromes, chronic liver disease, rheumatoid arthritis).
* Knowingly affected by HIV or viral hepatitis.
* History of local radiation therapy in the last five years.
* Affected by limited mental capacity or language skills such that study information cannot be understood, informed consent cannot be obtained, or simple instructions cannot be followed.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality which may increase the risk associated with trial participation or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this trial.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Women in menopause
Study Population: All post-menopausal women ≥ 65 years old attending the Centro Universitario di Odontoiatria in the new patients' or follow-ups' clinics will be approached to check for the inclusion/exclusion criteria and their willingness to take part in the study. Furthermore, doctors (general practitioners or osteoporosis specialists) will be contacted and will be kindly asked to inform their patient that had done a DXA scan within the past 12 months about the study. Potentially eligible patients will be booked an appointment at the "Centro Universitario di Odontoiatria, Dipartimento di Medicina e Chirurgia, Università di Parma" to check for inclusion/exclusion criteria and for the recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
sensitivity and specificity of Klemetti Index | 12 months is the maximum time between DXA results and OPT results, so it is also the timing for this outcome measurement
  To assess the sensitivity and specificity of Klemetti Index (KI) to screen for osteoporosis in postmenopausal women attending the Centre of Dentistry at the University of Parma

SECONDARY OUTCOMES:
sensitivity and specificity of mandibular cortical width | 12 months is the maximum time between DXA results and OPT results, so it is also the timing for this outcome measurement
  To assess the sensitivity and specificity of mandibular cortical width (MCW) to screen for osteoporosis in postmenopausal women
sensitivity and specificity of panoramic mandibular index | 12 months is the maximum time between DXA results and OPT results, so it is also the timing for this outcome measurement
  To assess the sensitivity and specificity of panoramic mandibular index (PMI) to screen for osteoporosis in postmenopausal women
Precision and reproducibility of Klemetti index | 12 months is the maximum time between DXA results and OPT results, so it is also the timing for this outcome measurement
  Two blind examiners will calculate the index twice (within at least one week from the first evaluation) and intra and inter examiner reproducibility will be assessed through Kappa statistics
Number of post-menopausal women attending a University Dental Hospital (Centro Universitario di Odontoiatria) and identified as osteoporotic with the help of the panoramic indices | up to 18 months
number of osteoporotic women identified as osteoporotic with the help of panoramic indices and their risk of fractures | At study completion, up to 18 months from the beginning of the study
  this will be calculated based on the Italian modified version of FRAX, "DeFRA"

CONTACTS AND LOCATIONS:
Overall Officials: Elena Calciolari, DDS, MS, PHD, Principal Investigator — University of Parma and Queen Mary University of London
Locations (1):
- Centro Universitario di Odontoiatria, Parma, Italy

IPD SHARING:
Plan to Share IPD: No
Information with regards to study participants will be kept confidential and data will be pseudo anonymised

REFERENCES:
- [Background] Calciolari E, Donos N, Park JC, Petrie A, Mardas N. Panoramic measures for oral bone mass in detecting osteoporosis: a systematic review and meta-analysis. J Dent Res. 2015 Mar;94(3 Suppl):17S-27S. doi: 10.1177/0022034514554949. Epub 2014 Nov 3. PMID 25365969
- [Background] Calciolari E, Donos N, Park JC, Petrie A, Mardas N. A systematic review on the correlation between skeletal and jawbone mineral density in osteoporotic subjects. Clin Oral Implants Res. 2016 Apr;27(4):433-42. doi: 10.1111/clr.12597. Epub 2015 Apr 12. PMID 25864584
- [Background] Klemetti E, Kolmakov S, Kroger H. Pantomography in assessment of the osteoporosis risk group. Scand J Dent Res. 1994 Feb;102(1):68-72. doi: 10.1111/j.1600-0722.1994.tb01156.x. PMID 8153584
- [Background] Benson BW, Prihoda TJ, Glass BJ. Variations in adult cortical bone mass as measured by a panoramic mandibular index. Oral Surg Oral Med Oral Pathol. 1991 Mar;71(3):349-56. doi: 10.1016/0030-4220(91)90314-3. PMID 2011361
- [Background] Kanis JA, McCloskey EV, Johansson H, Cooper C, Rizzoli R, Reginster JY; Scientific Advisory Board of the European Society for Clinical and Economic Aspects of Osteoporosis and Osteoarthritis (ESCEO) and the Committee of Scientific Advisors of the International Osteoporosis Foundation (IOF). European guidance for the diagnosis and management of osteoporosis in postmenopausal women. Osteoporos Int. 2013 Jan;24(1):23-57. doi: 10.1007/s00198-012-2074-y. Epub 2012 Oct 19. PMID 23079689
- [Background] Horner K, Devlin H. The relationship between mandibular bone mineral density and panoramic radiographic measurements. J Dent. 1998 May;26(4):337-43. doi: 10.1016/s0300-5712(97)00020-1. PMID 9611939